CLINICAL TRIAL: NCT01541072
Title: Lymphocyte Reconstitution in a Randomized Study After Administration of Pegfilgrastim Versus Filgrastim in Patients With B-cell Non-Hodgkin Lymphoma Treated With High-dose Chemotherapy and Autologous Peripheral Stem Cell Transplantation
Brief Title: Lymphocyte Reconstitution After Administration of Pegfilgrastim Versus Filgrastim After Peripheral Stem Cell Transplantation
Acronym: PALM2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Number of enrolled patients was insufficient during planned inclusion time.
Sponsor: Centre Leon Berard (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ET2011-010; 2011-A00662-39 (Registry Identifier: RCB)
Record Dates: First submitted 2012-02-17; First posted 2012-02-29 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Non Hodgkin Lymphoma
Keywords: Lymphoma, B-cell; Lymphocyte reconstitution; Lymphocyte subsets; Peripheral stem cell transplantation; Induction chemotherapy; growth factor; Granulocyte Colony-stimulating factor; Pegfilgrastim; Filgrastim
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell | interventions — pegfilgrastim; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pegfilgrastim (Experimental)
  Interventions: Drug: Pegfilgrastim
- Filgrastim (Active Comparator)
  Interventions: Drug: Filgrastim

INTERVENTIONS:
Drug: Pegfilgrastim — Pegfilgrastim (Neulasta®, AMGEN Laboratories): single subcutaneous administration of Pegfilgrastim, 6 mg at day 5 (D5) after autologous stem cell transplantation
  Other Names: Neulasta, AMGEN Laboratories
  Arms: Pegfilgrastim
Drug: Filgrastim — Filgrastim (Neupogen®, AMGEN Laboratories): daily subcutaneous administration, 5µg/kg/day from day 5 (D5) after autologous stem cell transplantation until recovery from aplasia (Neutrophils >= 0.5 G/L)
  Other Names: Neupogen, AMGEN Laboratories
  Arms: Filgrastim

SUMMARY:
The purpose of this study is to describe the kinetics of lymphocyte subsets reconstitution after growth factor administration, Pegfilgrastim versus Filgrastim in patients with B-cell malignant non-Hodgkin lymphoma treated with high-dose chemotherapy and autologous peripheral stem cell transplantation.

DETAILED DESCRIPTION:
High dose chemotherapy with autologous peripheral stem cell transplantation is a standard consolidation treatment used in patients with non-Hodgkin lymphoma, in first or second line of treatment. This procedure is associated with prolonged neutropenia and considerable morbidity. Different guidelines have recommended the use of growth factor after peripheral stem cell transplantation.Pegfilgrastim is a granulocyte colony-stimulating factor (G-CSF) resulting from the modification of Filgrastim by chemical addition of a polyethylene glycol(PEG) moiety which increases its half-life by decreasing its renal clearance. Then, a single injection substitutes several Filgrastim injections. The trial "PALM" realized by our team has shown, between these 2 molecules, an equivalent efficacy on the duration of chemotherapy-induced febrile neutropenia in patients treated for lymphoma or myeloma. This trial has also shown that Pegfilgrastim is a cost-effectiveness dominant strategy.

Some studies have shown that a rapid lymphocyte reconstitution after stem cell transplantation is associated with better overall survival and progression-free survival.

In the present PALM2 study, the investigators want to describe the kinetics of different lymphocyte subsets reconstitution within 3 and 6 months after transplantation, in patients with B-cell malignant non-Hodgkin lymphoma, in first or second-line chemotherapy and first autologous transplantation. The investigators will assess the kinetics of reconstitution for T-lymphocytes (Naïve T-lymphocytes, regulatory T-cells and memory T-cells), B-lymphocytes (transitional B cells), cytotoxic T-cells and natural killer T-cells, dendritic cells. A preliminary phase to this assessment will consist in estimate intra-center variability of lymphocyte phenotyping.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patients with B-cell NHL, except Burkitt Lymphoma and primary brain lymphoma, as first-line or second-line therapy, with planed BICNU, etoposide, aracytine and melphalan (BEAM) chemotherapy after pre-inclusion.
* Minimum one mobilization with G-CSF, G-CSF and endoxan or mozobil
* Minimum one cytapheresis with CD34>2 millions CD34/kg for stem cell transplantation
* Patients hospitalized in the investigational center throughout the procedure and until recovery from aplasia (neutrophils> 0.5 G/L)
* Mandatory affiliation with a health insurance system
* Subjects must provide written informed consent prior to performance of study-specific assessments

Exclusion Criteria:

* Patients already treated with intensive chemotherapy and autologous stem cell transplantation
* Total irradiation exposure (patients with partial irradiation exposure can be included in the study)
* Intolerance to one of the two studied growth factors, or hypersensitivity to one of their components
* Patients with neutropenia (neutrophils <1.2 G/L) or thrombopenia (platelets < 100 G/L) before intensive chemotherapy
* Acquired immune deficiency syndrome, seropositivity
* Pregnant or lactating women (pregnancy test, for women of childbearing potential, should be negative, in blood or urine, at inclusion time)
* Impossibility to comply with protocol constraints because of geographical, psychiatric, social or family reasons
* Deprived of liberty (court judgement or administrative decision)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-02; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
3 months kinetics of lymphocyte reconstitution, in the two arms | Lymphocyte count within the 3 months post transplantation

SECONDARY OUTCOMES:
6 months kinetics of lymphocyte reconstitution, in the two arms | Lymphocyte count within the 6 months post transplantation
6 months kinetics of lymphocyte subsets reconstitution by phenotyping, in the 2 arms | In the transplant and within the 6 months after transplantation (at Day 15, D30, D90, D180 after transplantation)
Average duration of neutropenia and thrombopenia, in the 2 arms | Within the 3 months post transplantation
  1. neutrophils<0.5 G/L
  2. neutrophils<1 G/L
  3. platelets<20 G/L
  4. platelets<50 G/L
Number of days with temperature ≥38°, in the 2 arms | For duration of post transplantation hospital stay, an expected average of 2 weeks
Number of bacterial and/or viral and/or fungal infection longer than 7 days, average duration of anti-viral, anti-fungal and antibiotic treatments, in the 2 arms | Within 3 months post transplantation
Number of red blood cell units and platelets concentrates transfused to patient, in the 2 arms | Within 3 months post transplantation
Evaluation of duration of Filgrastim treatment, in arm "Filgrastim" | For duration of post transplantation hospital stay, an expected average of 2 weeks
Overall survival | Within 18 months after the first inclusion, from the date of randomization until the date of death from any cause
Progression free survival | Within 18 months after yhe first inclusion, from the date of randomization until the date of the first documented progression or death from any cause, whichever came first
  The progression is measured as per 2007 Cheson international response criteria. Cheson BD et al. Revised response criteria for malignant lymphoma. J of Clin Oncol 2007;25(5):579-586
Average duration of febrile neutropenia (with neutrophils<0.5 G/L and temperature ≥38°), in the 2 arms | For duration of post transplantation hospital stay, an expected duration of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Catherine SEBBAN, MD, Principal Investigator — Centre Leon Berard, Lyon, France
Locations (2):
- France (2):
  - CHU Clermont-Ferrand, Hôpital d'Estaing, Clermont-Ferrand
  - Centre Leon Berard, Lyon

REFERENCES:
- [Background] Dieckmann D, Plottner H, Berchtold S, Berger T, Schuler G. Ex vivo isolation and characterization of CD4(+)CD25(+) T cells with regulatory properties from human blood. J Exp Med. 2001 Jun 4;193(11):1303-10. doi: 10.1084/jem.193.11.1303. PMID 11390437
- [Background] Goguel AF, Crainic K, Ducailar A, Ouin M. Interlaboratory quality assessment of lymphocyte phenotyping. Etalonorme 1990-1992 surveys. Biol Cell. 1993;78(1-2):79-84. doi: 10.1016/0248-4900(93)90118-x. PMID 8220229
- [Background] Holmes FA, Jones SE, O'Shaughnessy J, Vukelja S, George T, Savin M, Richards D, Glaspy J, Meza L, Cohen G, Dhami M, Budman DR, Hackett J, Brassard M, Yang BB, Liang BC. Comparable efficacy and safety profiles of once-per-cycle pegfilgrastim and daily injection filgrastim in chemotherapy-induced neutropenia: a multicenter dose-finding study in women with breast cancer. Ann Oncol. 2002 Jun;13(6):903-9. doi: 10.1093/annonc/mdf130. PMID 12123336
- [Background] Holmes FA, O'Shaughnessy JA, Vukelja S, Jones SE, Shogan J, Savin M, Glaspy J, Moore M, Meza L, Wiznitzer I, Neumann TA, Hill LR, Liang BC. Blinded, randomized, multicenter study to evaluate single administration pegfilgrastim once per cycle versus daily filgrastim as an adjunct to chemotherapy in patients with high-risk stage II or stage III/IV breast cancer. J Clin Oncol. 2002 Feb 1;20(3):727-31. doi: 10.1200/JCO.2002.20.3.727. PMID 11821454
- [Background] Joao C, Porrata LF, Inwards DJ, Ansell SM, Micallef IN, Johnston PB, Gastineau DA, Markovic SN. Early lymphocyte recovery after autologous stem cell transplantation predicts superior survival in mantle-cell lymphoma. Bone Marrow Transplant. 2006 May;37(9):865-71. doi: 10.1038/sj.bmt.1705342. PMID 16532015
- [Background] Jonuleit H, Schmitt E, Stassen M, Tuettenberg A, Knop J, Enk AH. Identification and functional characterization of human CD4(+)CD25(+) T cells with regulatory properties isolated from peripheral blood. J Exp Med. 2001 Jun 4;193(11):1285-94. doi: 10.1084/jem.193.11.1285. PMID 11390435
- [Background] Noether, G. E. Sample size determination for some common nonparametric statistics. Journal of the American Statistical Association 82 : 645-47, 1987.
- [Background] Peggs KS. Immune reconstitution following stem cell transplantation. Leuk Lymphoma. 2004 Jun;45(6):1093-101. doi: 10.1080/10428190310001641260. PMID 15359987
- [Background] Porrata LF, Gertz MA, Inwards DJ, Litzow MR, Lacy MQ, Tefferi A, Gastineau DA, Dispenzieri A, Ansell SM, Micallef IN, Geyer SM, Markovic SN. Early lymphocyte recovery predicts superior survival after autologous hematopoietic stem cell transplantation in multiple myeloma or non-Hodgkin lymphoma. Blood. 2001 Aug 1;98(3):579-85. doi: 10.1182/blood.v98.3.579. PMID 11468153
- [Background] Porrata LF, Inwards DJ, Ansell SM, Micallef IN, Johnston PB, Gastineau DA, Litzow MR, Winters JL, Markovic SN. Early lymphocyte recovery predicts superior survival after autologous stem cell transplantation in non-Hodgkin lymphoma: a prospective study. Biol Blood Marrow Transplant. 2008 Jul;14(7):807-16. doi: 10.1016/j.bbmt.2008.04.013. PMID 18541201
- [Background] Porrata LF, Inwards DJ, Micallef IN, Ansell SM, Geyer SM, Markovic SN. Early lymphocyte recovery post-autologous haematopoietic stem cell transplantation is associated with better survival in Hodgkin's disease. Br J Haematol. 2002 Jun;117(3):629-33. doi: 10.1046/j.1365-2141.2002.03478.x. PMID 12028034
- [Background] Reimer P, Kunzmann V, Wilhelm M, Weissbrich B, Kraemer D, Berghammer H, Weissinger F. Cellular and humoral immune reconstitution after autologous peripheral blood stem cell transplantation (PBSCT). Ann Hematol. 2003 May;82(5):263-70. doi: 10.1007/s00277-003-0630-4. Epub 2003 Mar 22. PMID 12739062
- [Background] Roberts MM, To LB, Gillis D, Mundy J, Rawling C, Ng K, Juttner CA. Immune reconstitution following peripheral blood stem cell transplantation, autologous bone marrow transplantation and allogeneic bone marrow transplantation. Bone Marrow Transplant. 1993 Nov;12(5):469-75. PMID 7905331
- [Background] Sebban, C., Lefranc, A, Perrier, L., Morreau, P., Espinouse, D., Moles-Moreau, M-P, Kammoun, L, Ghesquieres, H, Segura-Ferlay, C., Bay, J-O, Lissandre, S, PEROL, D, Michallet, M, and Quittet, P. A Randomized Phase II Study Evaluating the Efficacy, Safety and Cost-Effectiveness of Pegfilgrastim and Filgrastim After High Dose Chemotherapy and Autologous Stem Cell Transplantation In Patients with Lymphoma and Myeloma (PALM Study). ASH . 4-12-2010. Ref Type: Abstract
- [Background] Shimizu J, Yamazaki S, Sakaguchi S. Induction of tumor immunity by removing CD25+CD4+ T cells: a common basis between tumor immunity and autoimmunity. J Immunol. 1999 Nov 15;163(10):5211-8. PMID 10553041
- [Background] Singh RK, Ino K, Varney ML, Heimann DG, Talmadge JE. Immunoregulatory cytokines in bone marrow and peripheral blood stem cell products. Bone Marrow Transplant. 1999 Jan;23(1):53-62. doi: 10.1038/sj.bmt.1701518. PMID 10037051
- [Background] Talmadge JE, Reed E, Ino K, Kessinger A, Kuszynski C, Heimann D, Varney M, Jackson J, Vose JM, Bierman PJ. Rapid immunologic reconstitution following transplantation with mobilized peripheral blood stem cells as compared to bone marrow. Bone Marrow Transplant. 1997 Jan;19(2):161-72. doi: 10.1038/sj.bmt.1700626. PMID 9116614
- [Background] Thornton AM, Shevach EM. Suppressor effector function of CD4+CD25+ immunoregulatory T cells is antigen nonspecific. J Immunol. 2000 Jan 1;164(1):183-90. doi: 10.4049/jimmunol.164.1.183. PMID 10605010
- [Background] Vanstraelen G, Frere P, Ngirabacu MC, Willems E, Fillet G, Beguin Y. Pegfilgrastim compared with Filgrastim after autologous hematopoietic peripheral blood stem cell transplantation. Exp Hematol. 2006 Mar;34(3):382-8. doi: 10.1016/j.exphem.2005.11.013. PMID 16543072
- [Background] Woo EY, Chu CS, Goletz TJ, Schlienger K, Yeh H, Coukos G, Rubin SC, Kaiser LR, June CH. Regulatory CD4(+)CD25(+) T cells in tumors from patients with early-stage non-small cell lung cancer and late-stage ovarian cancer. Cancer Res. 2001 Jun 15;61(12):4766-72. PMID 11406550